CLINICAL TRIAL: NCT02471144
Title: A Randomized, Double-blind, Placebo- and Active Controlled Multicenter Trial to Demonstrate Efficacy of Subcutaneous Secukinumab Compared to Placebo and Etanercept (in a Single-blinded Arm) After Twelve Weeks of Treatment, and to Assess the Safety, Tolerability, and Long-term Efficacy in Subjects From 6 to Less Than 18 Years of Age With Severe Chronic Plaque Psoriasis
Brief Title: Pediatric Study in Children and Adolescents With Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2310; 2014-005663-32 (EudraCT Number)
Record Dates: First submitted 2015-05-04; First posted 2015-06-15 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Chronic Severe Plaque-type Psoriasis
Keywords: pediatric; chronic severe plaque psoriasis; secukinumab; etanercept
MeSH Terms: interventions — secukinumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Secukinumab low dose (Experimental): Secukinumab
  Interventions: Biological: Experimental : Secukinumab low dose
- Secukinumab high dose (Experimental): Secukinumab
  Interventions: Biological: Experimental: Secukinumab high dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo Comparator: Secukinumab Placebo
- Etanercept Comparator (Active Comparator): Etanercept
  Interventions: Biological: Active Comparator: Etanercept

INTERVENTIONS:
Biological: Experimental : Secukinumab low dose — Depending on weight group subject will receive per dose a) 75 mg if weighing less than 50 kg b) 150 mg if weighing 50 kg or more. Secukinumab injections (one or two per dose, depending on the weight group) will be administered subcutaneously at Randomization, Weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48, and Placebo secukinumab at Weeks 13, 14 and 15 during the blinded phase of the study; thereafter at Week 52 and every 4 weeks during the extension treatment period until Week 232.
  Other Names: AIN457 low dose
  Arms: Secukinumab low dose
Biological: Experimental: Secukinumab high dose — Depending on weight group subject will receive per dose a) 75 mg if weighing less than 25 kg b) 150 mg if weighing between 25 and less than 50 kg c) 300 mg if weighing more than 50 kg. Secukinumab injections (one or two per dose, depending on the weight group) will be administered subcutaneously at Randomization, Weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48, and Placebo secukinumab at Weeks 13, 14 and 15 during the blinded phase of the study; thereafter at Week 52 and every 4 weeks during the extension treatment period until Week 232.
  Other Names: AIN457 high dose
  Arms: Secukinumab high dose
Biological: Placebo Comparator: Secukinumab Placebo — Placebo secukinumab (one or two subcutaneous injections per dose, depending on weight group) at Randomization and Weeks 1, 2, 3 4 and 8. At Week 12, subjects in the placebo group based on their PASI 75 response status at Week 12 will proceed as follows: • PASI 75 responders will discontinue study treatment at Week 12 and enter the treatment-free follow-up period • PASI 75 non-responders will receive high dose or low dose secukinumab, according to the pre-assignment at the Randomization visit. They will receive their treatment based on the weight category(<25 kg, 25- <50kg, ≥50 kg), on Weeks 12, 13, 14, 15, and then every four weeks starting at Week 16 until Week 48 during the maintenance period; thereafter at week 52 and every 4 weeks during the extension treatment period until Week 232.
  Other Names: AIN457 placebo
  Arms: Placebo
Biological: Active Comparator: Etanercept — Etanercept 0.8 mg/kg of subject weight and up to a maximum of 50 mg per dose. Subcutaneous etanercept 0.8 mg/kg (one or two injections per dose) once per week, for 51 weeks administered at home (self-injected or by caregiver) or at the study site. At Wk 52 subjects in the etanercept group will move into the treatment-free follow up period and terminate the study.
  Other Names: Etanercept
  Arms: Etanercept Comparator

SUMMARY:
This was a multicenter, randomized, double-blind, placebo- and active-controlled (etanercept in single blinded arm) study in pediatric subjects aged 6 years to less than 18 years with severe chronic plaque psoriasis. Approximately 160 subjects aged 6 years to <18 years were enrolled, of which at least 30 were 6 years to <12 years old. Subjects were enrolled at approximately 70 study sites worldwide.

DETAILED DESCRIPTION:
The purpose of this study was to demonstrate superior efficacy of secukinumab versus placebo at Week 12, based on both PASI 75 and IGA mod 2011 0 or 1 response rates in children and adolescents aged 6 to less than 18 years with severe chronic plaque psoriasis who had inadequate control of symptoms with topical treatment, or failed to respond to or tolerate previous systemic treatment and/or UV therapy

The study assessed the long term safety and tolerability of secukinumab in this pediatric age group and described the efficacy and safety of secukinumab compared to etanercept. This study provided efficacy and safety data to support the extension of label of secukinumab to include children and adolescents (6 years to <18 years) with severe chronic plaque psoriasis

Two age subgroups were studied in a staggered approach within this clinical study: 12 to less than 18 years of age, and 6 to less than 12 years of age . Enrolment of children aged 6 to less than 12 years began after a favorable recommendation by an independent external Data Monitoring Committee (DMC) who reviewed data of approximately 80 adolescents. Adolescents continued to be recruited while the data from the first 80 subjects was being collected and analyzed

Subjects were randomized using a 1:1:1:1 ratio into one of the treatment arms: secukinumab low dose, secukinumab high dose, etanercept or placebo. Subjects randomized to secukinumab treatment arms (high dose and low dose) received dose based on the weight category (<25 kg, 25 to <50kg, ≥50 kg).

The study consisted of 5 periods: screening (up to 4 weeks), induction (of 12 weeks), maintenance (of 40 weeks), extension treatment epoch (open-label of 184 weeks) and post- treatment follow-up epoch (of 16 weeks).

The screening period of up to 4 weeks was used to assess eligibility of the patients and to taper patients off prohibited medications.

The Induction period is defined as randomization through Week 12. In this period, the study was both active and placebo-controlled and at its completion, the primary endpoint was assessed (Week 12).

The Maintenance period is defined as Week 12 (from dosing) through Week 52. During this period, the study was active-controlled, and the objectives focused on the maintenance of the response observed at Week 12.

Patients who received secukinumab or etanercept during induction continued in maintenance with the same treatment. Patients who were on placebo during induction and at Week 12 were PASI 75 non-responders were switched to either secukinumab low dose or secukinumab high dose treatment group in the Maintenance period according to their baseline randomization.

At the end of the Maintenance period, all patients on secukinumab entered the Extension treatment period and continued to receive the same dose of secukinumab. The Extension treatment period was defined as Week 52 (from dosing) until Week 236. In this period, all patients were treated with secukinumab, and the purpose was the collection of long-term safety and efficacy data.

Patients who participated in the Maintenance period but prematurely discontinued the study were not able to enter the Extension treatment period. Patients receiving etanercept were not eligible to enter the Extension treatment period. Instead, at Week 52, they completed an EOM visit and then entered the post-treatment Follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Must be 6 to less than 18 years of age at the time of randomization
* Plaque-type psoriasis history for at least 3 months.

Severe plaque-type psoriasis meeting all of the following three criteria:

* PASI score of 20 or greater,
* Investigator's Global Assessment (IGA) score of 4
* Total body surface area (BSA) affected of 10% or greater.
* Patient being regarded by the investigator to be a candidate for systemic therapy because of:

  1. inadequate control of symptoms with topical treatment, or
  2. failure to respond to or tolerate previous systemic treatment and/or UV therapy

Exclusion criteria

* Current forms of psoriasis other than chronic plaque-type psoriasis (for example, pustular, erythrodermic, guttate) at randomization.
* Current drug-induced psoriasis.
* Previous use of secukinumab or any drug that targets IL-17 or IL-17 receptor.
* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy
* History of an ongoing, chronic or recurrent infectious disease, or evidence of untreated tuberculosis.
* History of lymphoproliferative disease or history of malignancy of any organ system within the past 5 years.
* Pregnant or nursing (lactating) women.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- Novartis Investigative Site, San Antonio, Texas, United States
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogotá
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- Novartis Investigative Site, Tartu, Estonia
- France (3):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Ramat Gan
- Italy (2):
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Nagoya, Aichi-ken, Japan
- Novartis Investigative Site, Riga, Latvia
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Cluj-Napoca, Cluj, Romania
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Spain (3):
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Scunthorpe, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sticherling M, Nikkels AF, Hamza AM, Kwong P, Szepietowski JC, El Sayed M, Ghislain PD, Khotko AA, Patekar M, Ortmann CE, Forrer P, Papanastasiou P, Keefe D. Secukinumab in Pediatric Patients with Plaque Psoriasis: Pooled Safety Analysis from Two Phase 3 Randomized Clinical Trials. Am J Clin Dermatol. 2023 Sep;24(5):821-835. doi: 10.1007/s40257-023-00782-8. Epub 2023 Jun 21. PMID 37341961
- [Derived] Krasowska D, Gambichler T, Cortes C, Horev A, Compagno N, Dahale SS, Papanastasiou P, Keefe D. Long-term efficacy, safety and tolerability of secukinumab in children and adolescents with severe chronic plaque psoriasis: Two-year results from a Phase III double-blind, randomized controlled trial. J Eur Acad Dermatol Venereol. 2023 Mar 27. doi: 10.1111/jdv.19063. Online ahead of print. PMID 36971771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-blind, placebo- and active-controlled (etanercept in single blinded arm) study in pediatric patients aged 6 years to less than 18 years with severe chronic plaque psoriasis. A total of 187 patients were screened, of which 162 were randomized.
Groups:
- AIN457 Low Dose (Induction Period); AIN457 Low Dose (Maintenance Period): Patients received secukinumab 75mg (if weighing < 50kg) or 150 mg (if weighing >=50 kg) at each dosing
- AIN457 High Dose (Induction Period); AIN457 High Dose (Maintenance Period): Patients received secukinumab 75mg (if weighing < 25kg) or 150 mg (if weighing 25 to < 50kg ) or 300 mg (if weighing >=50 kg) at each dosing
- Placebo (Induction Period): Patients received matching placebo to secukinumab at each dosing
- Etanercept Comparator (Induction Period); Etanercept Comparator (Maintenance Period): Patients received weekly open label etanercept 0.8 mg/kg of body weight (up to a maximum of 50 mg)
- Placebo-AIN457 Low Dose (Maintenance Period): Patients received placebo during Induction and if they were PASI 75 non-responders at Week 12 switched to AIN457 Low Dose for the remainder of the study
- Placebo-AIN457 High Dose (Maintenance Period: Patients received placebo during Induction and if they were PASI 75 non-responders at Week 12 switched to AIN457 High Dose for the remainder of the study
- Any AIN457 Low Dose (Extension Period): Includes patients from the AIN457 Low Dose and from the Placebo-AIN457 Low Dose groups
- Any AIN457 High Dose (Extension Period): Includes patients from the AIN457 High Dose and from the Placebo-AIN457 High Dose groups
Period: Induction Period (Up to Week 12)
Arm/Group | AIN457 Low Dose (Induction Period) | AIN457 High Dose (Induction Period) | Placebo (Induction Period) | Etanercept Comparator (Induction Period) | AIN457 Low Dose (Maintenance Period) | AIN457 High Dose (Maintenance Period) | Placebo-AIN457 Low Dose (Maintenance Period) | Placebo-AIN457 High Dose (Maintenance Period | Etanercept Comparator (Maintenance Period) | Any AIN457 Low Dose (Extension Period) | Any AIN457 High Dose (Extension Period)
Started | 40 | 40 | 41 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 39 | 38 | 39 | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject/Guardian Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 12 to Week 52)
Arm/Group | AIN457 Low Dose (Induction Period) | AIN457 High Dose (Induction Period) | Placebo (Induction Period) | Etanercept Comparator (Induction Period) | AIN457 Low Dose (Maintenance Period) | AIN457 High Dose (Maintenance Period) | Placebo-AIN457 Low Dose (Maintenance Period) | Placebo-AIN457 High Dose (Maintenance Period | Etanercept Comparator (Maintenance Period) | Any AIN457 Low Dose (Extension Period) | Any AIN457 High Dose (Extension Period)
Started | 0 | 0 | 0 | 0 | 39 | 38 | 16 | 18 | 40 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 38 | 37 | 15 | 16 | 34 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 6 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Period: Extension Period (Week 52 to Week 236)
Arm/Group | AIN457 Low Dose (Induction Period) | AIN457 High Dose (Induction Period) | Placebo (Induction Period) | Etanercept Comparator (Induction Period) | AIN457 Low Dose (Maintenance Period) | AIN457 High Dose (Maintenance Period) | Placebo-AIN457 Low Dose (Maintenance Period) | Placebo-AIN457 High Dose (Maintenance Period | Etanercept Comparator (Maintenance Period) | Any AIN457 Low Dose (Extension Period) | Any AIN457 High Dose (Extension Period)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 53
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 43
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 10
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Technical problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: The randomized set was defined as all patients who were randomized. Mis-randomized patients were excluded from the randomized set. If patients were re screened and successfully randomized, they were included in the randomized set according to the treatment assigned in the last randomization.
Groups:
- AIN457 Low Dose: Patients received secukinumab 75mg (if weighing < 50kg) or 150 mg (if weighing >=50 kg) at each dosing
- AIN457 High Dose: Patients received secukinumab 75mg (if weighing < 25kg) or 150 mg (if weighing 25 to < 50kg ) or 300 mg (if weighing >=50 kg) at each dosing
- Placebo: Patients received matching placebo to secukinumab at each dosing
- Etanercept: Patients received weekly open label etanercept 0.8 mg/kg of body weight (up to a maximum of 50 mg)
- Total: Total of all reporting groups
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept | Total
Number analyzed (Participants) | 40 | 40 | 41 | 41 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.7 (2.92) | 13.2 (3.21) | 13.7 (3.27) | 13.5 (2.94) | 13.5 (3.06)
Age, Customized [Number; unit: Participants] — Age Categorical
  Participants
    <12 years | 8 | 9 | 10 | 10 | 37
    >=12 years | 32 | 31 | 31 | 31 | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 22 | 25 | 97
  Male | 13 | 17 | 19 | 16 | 65
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 34 | 34 | 36 | 30 | 134
  Black | 1 | 1 | 0 | 0 | 2
  Asian | 1 | 2 | 1 | 3 | 7
  Native American | 3 | 3 | 3 | 8 | 17
  Other | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Achieving a 75% Improvement From Baseline in PASI Score at Week 12
Description: Psoriasis Area and Severity Index (PASI):Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs and lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, Erythema,Thickening (plaque elevation, induration) & Scaling(desquamation). Scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, upper limbs: 0.2 trunk: 0.3 lower limbs: 0.4). Psoriasis Area and Severity Index (PASI) will be assessed/calculated as per standard procedure. PASI 75 represents the percentage (or number) of patients who have achieved a 75% or more reduction in their PASI score from baseline.
Time Frame: 12 weeks
Population: Full Analysis Set: The FAS comprised all patients from the randomized set to whom study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned at randomization. If the actual stratum was different to the assigned stratum in Interactive Response Technology (IRT), the actual stratum was used in analyses. Patients excluded from the randomized set were excluded from the FAS
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 41 | 41
Participants | 32 | 31 | 6 | 26
Statistical Analysis 1: Comparison: AIN457 Low Dose; vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 25.78, 95% CI 2-sided [7.08 to 114.66]
Statistical Analysis 2: Comparison: AIN457 High Dose; vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 22.65, 95% CI 2-sided [6.31 to 98.93]

2. Primary Outcome: Number and Percentage of Participants Who Showed Investigator's Global Assessment (IGA) Mod 2011 Response of 0 or 1 at Week 12
Description: IGA: The IGA mod 2011 scale has following different scores for the state of disease: 0: Clear, No signs of psoriasis. 1: Almost clear 2: Mild 3: Moderate 4 : Severe
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 40 | 41
Participants | 28 | 24 | 2 | 14
Statistical Analysis 1: Comparison: AIN457 Low Dose; vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 51.77, 95% CI 2-sided [10.02 to 538.64]
Statistical Analysis 2: Comparison: AIN457 High Dose; vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 32.52, 95% CI [6.48 to 329.52]

3. Secondary Outcome: Number and Percentage of Participants Achieving a 90% Improvement From Baseline in PASI Score at Week 12
Description: Psoriasis Area and Severity Index (PASI):Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs and lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, Erythema,Thickening (plaque elevation, induration) & Scaling(desquamation). Scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, upper limbs: 0.2 trunk: 0.3 lower limbs: 0.4). Psoriasis Area and Severity Index (PASI) will be assessed/calculated as per standard procedure. PASI 90 represents the percentage (or number) of patients who have achieved a 90% or more reduction in their PASI score from baseline.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 41 | 41
Participants | 29 | 27 | 1 | 12
Statistical Analysis 1: Comparison: AIN457 Low Dose; vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 72.5, 95% CI 2-sided [55.9 to 84.9]
Statistical Analysis 2: Comparison: AIN457 High Dose; vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 67.5, 95% CI 2-sided [50.8 to 80.9]

4. Secondary Outcome: Number and Percentage of Participants Achieving a 50%, 100% Improvement From Baseline in PASI Score at Week 12
Description: Psoriasis Area and Severity Index (PASI):Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs and lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, Erythema,Thickening (plaque elevation, induration) & Scaling(desquamation). Scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, upper limbs: 0.2 trunk: 0.3 lower limbs: 0.4). Psoriasis Area and Severity Index (PASI) will be assessed/calculated as per standard procedure. PASI 50 represents the percentage (or number) of patients who have achieved a 50% or more reduction in their PASI score from baseline. PASI 100 indicates patients who have achieved a complete resolution of all disease.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 41 | 41
Participants
  PASI 50 | 34 | 34 | 9 | 34
  PASI 100 | 12 | 11 | 0 | 7

5. Secondary Outcome: Number and Percentage of Participants Achieving a 50%, 75%, 90% or 100% Improvement From Baseline in PASI Score and IGA Mod 2011 Score of 0 or 1 up to Week 12 (Induction)
Description: Psoriasis Area and Severity Index (PASI):Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs and lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, Erythema, Thickening (plaque elevation, induration) & Scaling(desquamation). Scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, upper limbs: 0.2 trunk: 0.3 lower limbs: 0.4). PASI will be assessed/calculated as per standard procedure. IGA: The IGA mod 2011 scale has following different scores for the state of disease: 0: Clear, No signs of psoriasis. 1: Almost clear 2: Mild 3: Moderate 4 : Severe
Time Frame: Weeks 4, 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 41 | 41
Participants
  Week 4- IGA 0/1 | 6 | 13 | 0 | 1
  Week 4- PASI 50 | 26 | 28 | 6 | 19
  Week 4- PASI 75 | 13 | 22 | 0 | 5
  Week 4- PASI 90 | 5 | 9 | 0 | 1
  Week 4- PASI 100 | 3 | 3 | 0 | 0
  Week 8- IGA 0/1 | 21 | 18 | 0 | 6
  Week 8- PASI 50 | 32 | 32 | 11 | 30
  Week 8- PASI 75 | 27 | 26 | 1 | 15
  Week 8- PASI 90 | 20 | 20 | 0 | 4
  Week 8-PASI 100 | 9 | 7 | 0 | 2

6. Secondary Outcome: Number and Percentage of Participants Achieving a 50%, 75%, 90% or 100% Improvement From Baseline in PASI Score and IGA Mod 2011 Score of 0 or 1 Up to Week 52 (Maintenance)
Description: as for outcome 5
Time Frame: Weeks 16, 20, 24, 36, 48 and 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Placebo-AIN457 Low Dose: Patients received placebo during Induction and if they were PASI 75 non-responders at Week 12 switched to AIN457 Low Dose for the remainder of the study
- Placebo- AIN457 High Dose: Patients received placebo during Induction and if they were PASI 75 non-responders at Week 12 switched to AIN457 High Dose for the remainder of the study
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo-AIN457 Low Dose | Placebo- AIN457 High Dose | Etanercept
Number analyzed (Participants) | 40 | 40 | 16 | 18 | 41
Participants
  Week 16- IGA 0/1 | 32 | 28 | 5 | 8 | 19
  Week 16- PASI 50 | 37 | 35 | 11 | 16 | 30
  Week 16- PASI 75 | 36 | 32 | 5 | 11 | 26
  Week 16- PASI 90 | 33 | 30 | 4 | 7 | 16
  Week 16- PASI 100 | 19 | 14 | 0 | 1 | 8
  Week 20- IGA 0/1 | 33 | 28 | 12 | 13 | 21
  Week 20- PASI 50 | 38 | 36 | 15 | 17 | 32
  Week 20- PASI 75 | 38 | 35 | 13 | 15 | 29
  Week 20- PASI 90 | 33 | 30 | 12 | 12 | 19
  Week 20- PASI 100 | 20 | 16 | 5 | 4 | 8
  Week 24- IGA 0/1 | 35 | 30 | 14 | 14 | 20
  Week 24- PASI 50 | 38 | 37 | 15 | 16 | 31
  Week 24- PASI 75 | 37 | 35 | 15 | 14 | 26
  Week 24- PASI 90 | 33 | 31 | 13 | 12 | 19
  Week 24- PASI 100 | 22 | 17 | 7 | 6 | 9
  Week 36- IGA 0/1 | 32 | 29 | 14 | 14 | 21
  Week 36- PASI 50 | 37 | 37 | 16 | 16 | 31
  Week 36- PASI 75 | 35 | 35 | 16 | 16 | 26
  Week 36-PASI 90 | 32 | 31 | 10 | 7 | 18
  Week 36-PASI 100 | 17 | 20 | 10 | 7 | 10
  Week 48- IGA 0/1 | 28 | 28 | 14 | 14 | 21
  Week 48-PASI 50 | 38 | 35 | 15 | 15 | 31
  Week 48- PASI 75 | 35 | 35 | 14 | 15 | 27
  Week 48- PASI 90 | 29 | 30 | 12 | 14 | 23
  Week 48- PASI 100 | 16 | 18 | 10 | 8 | 12
  Week 52- 1GA 0/1 | 29 | 30 | 14 | 13 | 23
  Week 52- PASI 50 | 39 | 37 | 15 | 17 | 32
  Week 52- PASI 75 | 35 | 35 | 14 | 17 | 28
  Week 52- PASI 90 | 30 | 32 | 13 | 14 | 21
  Week 52- PASI 100 | 16 | 19 | 10 | 10 | 9

7. Secondary Outcome: Change From Baseline in Psoriasis Area & Severity Index (PASI) Score at Week 12
Description: Psoriasis Area and Severity Index (PASI):Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs and lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, Erythema,Thickening (plaque elevation, induration) & Scaling(desquamation). Scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, upper limbs: 0.2 trunk: 0.3 lower limbs: 0.4). Psoriasis Area and Severity Index (PASI) will be assessed/calculated as per standard procedure. PASI 75 represents the percentage (or number)of patients who have achieved a 75% or more reduction in their PASI score from baseline. PASI 100 indicates patients who have achieved a complete resolution of all disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 39 | 39 | 40 | 41
Scores on a scale | -22.27 (8.518) | -22.67 (11.904) | -7.94 (9.396) | -20.91 (10.055)

8. Secondary Outcome: Change From Baseline in Psoriasis Area & Severity Index (PASI) Scores at Week 52
Description: as for outcome 7
Time Frame: Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo-AIN457 High Dose: Patients received placebo during Induction and if they were PASI 75 non-responders at Week 12 switched to AIN457 High Dose for the remainder of the study
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo-AIN457 Low Dose | Placebo-AIN457 High Dose | Etanercept
Number analyzed (Participants) | 39 | 39 | 16 | 18 | 41
Scores on a scale | -25.26 (7.150) | -25.75 (8.593) | -28.49 (7.984) | -24.69 (5.520) | -21.16 (11.779)

9. Secondary Outcome: Percentage of Participants in IGA Mod 2011 Score Categories at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 41 | 41
Participants
  Week 12- IGA Category: Clear | 12 | 11 | 0 | 7
  Week 12- IGA Category: Almost Clear | 14 | 13 | 2 | 7
  Week 12- IGA Category: Mild Disease | 8 | 7 | 4 | 18
  Week 12- IGA Category: Moderate Disease | 3 | 4 | 11 | 6
  Week 12- IGA Category: Severe Disease | 2 | 4 | 23 | 3

10. Secondary Outcome: Percentage of Participants in IGA Mod 2011 Score Categories at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo-AIN457 Low Dose | Placebo-AIN457 High Dose | Etanercept
Number analyzed (Participants) | 40 | 40 | 16 | 18 | 41
Participants
  Week 52- IGA Category: Clear: number analyzed (Participants) | 39 | 39 | 16 | 18 | 41
  Week 52- IGA Category: Clear | 16 | 20 | 10 | 10 | 9
  Week 52- IGA Category: Almost Clear: number analyzed (Participants) | 39 | 39 | 16 | 18 | 41
  Week 52- IGA Category: Almost Clear | 13 | 10 | 4 | 4 | 14
  Week 52- IGA Category: Mild Disease: number analyzed (Participants) | 39 | 39 | 16 | 18 | 41
  Week 52- IGA Category: Mild Disease | 7 | 4 | 2 | 4 | 9
  Week 52- IGA Category: Moderate Disease: number analyzed (Participants) | 39 | 39 | 16 | 18 | 41
  Week 52- IGA Category: Moderate Disease | 2 | 2 | 0 | 0 | 4
  Week 52- IGA Category: Severe Disease: number analyzed (Participants) | 39 | 39 | 16 | 18 | 41
  Week 52- IGA Category: Severe Disease | 1 | 3 | 0 | 0 | 5

11. Secondary Outcome: Percentage Change From Baseline in Children's Dermatology Life Quality Index (cDLQI) Score Up to Week 12 (Induction)
Description: The CDLQI measures functional disability of subjects with dermatological disorders who are less than 18 years of age and it has been utilized as a relevant clinical measure in atopic dermatitis, as well as other dermatitis clinical trials. The CDLQI is a simple, validated, self-administered 10-item questionnaire. The instrument contains six functional scales (i.e., symptoms and feeling, leisure, school or holidays, personal relationships, sleep and treatment). The questions are based on the preceding week to permit accurate recall. For the CDLQI, each question will be answered on a 4-point Likert scale scored from 0 to 3. Seven scores will be derived from the CDLQI: the total score of each of the six dimensions as well as the total score over all items. The higher the score, the more quality of life is impaired.
Time Frame: Weeks 4, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change of score
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 41 | 41
percentage change of score
  Week 4: number analyzed (Participants) | 36 | 35 | 37 | 36
  Week 4 | -47.71 (45.743) | -50.71 (37.003) | 1.67 (104.216) | -35.13 (56.832)
  Week 8: number analyzed (Participants) | 38 | 37 | 39 | 37
  Week 8 | -61.60 (54.371) | -66.97 (32.040) | -17.77 (66.451) | -42.73 (54.026)
  Week 12: number analyzed (Participants) | 37 | 37 | 39 | 37
  Week 12 | -67.43 (41.602) | -62.5 (50.08) | -18.48 (80.018) | -62.80 (34.419)

12. Secondary Outcome: Percentage Change From Baseline in Children's Dermatology Life Quality Index (cDLQI) Score Up to Week 52 (Maintenance)
Description: as for outcome 11
Time Frame: Weeks 24, 36, 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change of score
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo-AIN457 Low Dose | Placebo-AIN457 High Dose | Etanercept
Number analyzed (Participants) | 40 | 40 | 16 | 18 | 41
percentage change of score
  Week 24: number analyzed (Participants) | 32 | 33 | 14 | 14 | 35
  Week 24 | -73.7 (55.02) | -53.9 (74.63) | 40.3 (477.93) | -73.8 (53.09) | -55.0 (44.98)
  Week 36: number analyzed (Participants) | 32 | 32 | 13 | 12 | 33
  Week 36 | -79.0 (31.99) | -56.2 (107.65) | -89.5 (19.11) | -69.4 (46.46) | -47.7 (45.01)
  Week 52: number analyzed (Participants) | 32 | 32 | 13 | 13 | 32
  Week 52 | -80.9 (39.38) | -58.6 (77.56) | -89.0 (15.73) | -86.0 (23.19) | -53.4 (56.99)

13. Secondary Outcome: Number and Percentage of Participants Achieving a Children's DLQI Score of 0 or 1 Over Time up to Week 12 (Induction)
Description: as for outcome 11
Time Frame: Weeks 4, 8, 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 40 | 40 | 41 | 41
Participants
  Week 4: number analyzed (Participants) | 37 | 36 | 38 | 40
  Week 4 | 8 | 11 | 2 | 9
  Week 8: number analyzed (Participants) | 39 | 38 | 40 | 41
  Week 8 | 15 | 19 | 7 | 10
  Week 12: number analyzed (Participants) | 38 | 38 | 40 | 41
  Week 12 | 17 | 19 | 6 | 15

14. Secondary Outcome: Number and Percentage of Participants Achieving a Children's DLQI Score of 0 or 1 Over Time up to Week 52 (Maintenance)
Description: as for outcome 11
Time Frame: Weeks 24, 36, 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo-AIN457 Low Dose | Placebo-AIN457 High Dose | Etanercept
Number analyzed (Participants) | 40 | 40 | 16 | 18 | 41
Participants
  Week 24: number analyzed (Participants) | 33 | 34 | 15 | 14 | 39
  Week 24 | 19 | 17 | 8 | 9 | 17
  Week 36: number analyzed (Participants) | 33 | 33 | 14 | 12 | 37
  Week 36 | 21 | 21 | 9 | 8 | 12
  Week 52: number analyzed (Participants) | 33 | 33 | 14 | 13 | 36
  Week 52 | 20 | 22 | 8 | 11 | 16

15. Secondary Outcome: Number and Percentage of Participants With Clinically Important Reduction in Disability as Evaluated by CHAQ Questionnaire Over Time at Week 12
Description: The CHAQ questionnaire is only done for children who in addition to psoriasis are also suffering from psoriatic arthritis. The questionnaire is completed by parent or legal guardian. It consists of multiple choice items concerning difficulty in performing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and other "activities". The person completing the questionnaire chooses from four response categories, ranging from 'without any difficulty' to 'unable to do'. Additionally two visual analog scales (overall well-being and pain of patient) must be performed.
Time Frame: Week 12
Population: No summary statistics were derived for CHAQ, due to the low number of subjects (11) who completed the CHAQ questionnaire: 4 from secukinumab low dose group, 3 from etanercept group, 2 from placebo - secukinumab high dose group and 1 each from secukinumab high dose group and placebo - secukinumab low dose group. At Week 12 analysis visit, 4 patients achieved CHAQ response (2 each from secukinumab low dose and etanercept groups)
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo | Etanercept
Number analyzed (Participants) | 4 | 2 | 2 | 3
Participants | 2 | 0 | 0 | 2

16. Secondary Outcome: Number and Percentage of Participants With Clinically Important Reduction in Disability as Evaluated by CHAQ Questionnaire Over Time at Week 52
Description: as for outcome 15
Time Frame: Week 52
Population: No summary statistics were derived for CHAQ, due to the low number of subjects (11) who completed the CHAQ questionnaire: 4 secukinumab low dose, 1 secukinumab high dose, 3 Etanercept, who were evaluable at Week 52 Visit. 5 patients achieved CHAQ response (2 from etanercept group, 2 from secukinumab low dose group and 1 from placebo - secukinumab low dose)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo- AIN457 Low Dose: Patients received placebo during Induction and if they were PASI 75 non-responders at Week 12 switched to AIN457 Low Dose for the remainder of the study
Arm/Group | AIN457 Low Dose | AIN457 High Dose | Placebo- AIN457 Low Dose | Placebo- AIN457 High Dose | Etanercept
Number analyzed (Participants) | 4 | 1 | 2 | 1 | 3
Participants | 2 | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study treatment until last dose of study treatment plus 16 weeks. In total 252 weeks for AIN457 arms and 68 weeks for Etanercept. Placebo PASI-75 responders at week 12 moved into the 16 weeks post-treatment follow-up. AEs were collected for 28 weeks. Placebo PASI-75 non-responders at week 12 switched to active AIN457 dose groups. AEs were collected for 12 weeks under Placebo and up to 240 weeks under AIN457 arms.
Description: Adverse Events are reported according to the actual treatment received at the onset of the AE.
Groups:
- Any AIN457 Low Dose: Includes patients from the AIN457 Low Dose and from the Placebo-AIN457 Low Dose groups.
  AEs were collected for up to 252 weeks.
- Any AIN457 High Dose: Includes patients from the AIN457 High Dose and from the Placebo-AIN457 High Dose groups.
  AEs were collected for up to 252 weeks.
- Any AIN457 Dose: Any AIN457 dose. AEs were collected for up to 252 weeks.
- Placebo: Patients received matching placebo to secukinumab at each dosing. AEs were collected for up to 28 weeks (12 weeks if participant switched to AIN457 at week 12).
- Etanercept: Patients received weekly open label etanercept 0.8 mg/kg of body weight (up to a maximum of 50 mg).
  AEs were collected for up to 68 weeks.
Arm/Group | Any AIN457 Low Dose | Any AIN457 High Dose | Any AIN457 Dose | Placebo | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/58 | 0/114 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 7/56 | 8/58 | 15/114 | 0/41 | 6/41
Other Adverse Events (participants affected / at risk) | 48/56 | 50/58 | 98/114 | 19/41 | 30/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 Low Dose (N=56) | Any AIN457 High Dose (N=58) | Any AIN457 Dose (N=114) | Placebo (N=41) | Etanercept (N=41)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pilonidal disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 Low Dose (N=56) | Any AIN457 High Dose (N=58) | Any AIN457 Dose (N=114) | Placebo (N=41) | Etanercept (N=41)
Eosinophilia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 4 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 6 | 10 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5 | 9 | 2 | 4
Dental caries (Gastrointestinal disorders) | 1 | 3 | 4 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 14 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 2 | 4
Toothache (Gastrointestinal disorders) | 1 | 4 | 5 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5 | 6 | 0 | 1
Asthenia (General disorders) | 1 | 3 | 4 | 1 | 0
Fatigue (General disorders) | 3 | 3 | 6 | 1 | 0
Pyrexia (General disorders) | 4 | 6 | 10 | 0 | 2
Bronchitis (Infections and infestations) | 3 | 6 | 9 | 2 | 3
COVID-19 (Infections and infestations) | 4 | 5 | 9 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 5 | 7 | 0 | 1
Folliculitis (Infections and infestations) | 3 | 4 | 7 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 3 | 8 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 3 | 1 | 4 | 1 | 2
Gastrointestinal infection (Infections and infestations) | 2 | 4 | 6 | 2 | 0
Impetigo (Infections and infestations) | 0 | 3 | 3 | 0 | 1
Influenza (Infections and infestations) | 4 | 0 | 4 | 3 | 3
Nasopharyngitis (Infections and infestations) | 17 | 25 | 42 | 1 | 11
Oral herpes (Infections and infestations) | 3 | 2 | 5 | 1 | 4
Paronychia (Infections and infestations) | 1 | 3 | 4 | 0 | 1
Pharyngitis (Infections and infestations) | 9 | 8 | 17 | 4 | 3
Pharyngotonsillitis (Infections and infestations) | 4 | 1 | 5 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 4 | 7 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 7 | 12 | 4 | 1
Sinusitis (Infections and infestations) | 4 | 2 | 6 | 0 | 1
Tonsillitis (Infections and infestations) | 11 | 7 | 18 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 3 | 10 | 3 | 3
Urinary tract infection (Infections and infestations) | 5 | 2 | 7 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 4 | 7 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 6 | 0 | 2
Glomerular filtration rate decreased (Investigations) | 7 | 4 | 11 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 9 | 1 | 2
Headache (Nervous system disorders) | 11 | 11 | 22 | 4 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 4 | 5 | 0 | 2
Menstruation irregular (Reproductive system and breast disorders) | 0 | 3 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 13 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 10 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 8 | 5 | 13 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 5 | 8 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 8 | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 7 | 1 | 8 | 0 | 4
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 4 | 6 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT02471144/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT02471144/SAP_001.pdf